CLINICAL TRIAL: NCT00515853
Title: The Role of Biofeedback in Improving Continence After Anterior Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHM GSU 0132
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-01

CONDITIONS: Rectal Neoplasms; Fecal Incontinence; Aged
Keywords: Rectal neoplasms; Biofeedback (Psychology); Fecal Incontinence; Aged; Anterior resection
MeSH Terms: conditions — Rectal Neoplasms; Fecal Incontinence | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): Received feedback
  Interventions: Behavioral: Biofeedback
- No biofeedback (No Intervention): Did not received feedback

INTERVENTIONS:
Behavioral: Biofeedback — Biofeedback sessions or biofeedback exercises
  Arms: Biofeedback

SUMMARY:
The purpose of this study is to determine whether biofeedback exercises improve anal continence after anterior resection for rectal cancer.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Rectosigmoid or rectal cancer

Exclusion Criteria:

* Inoperable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-11-27 (Actual); Primary Completion 2010-05-13 (Actual); Study Completion 2010-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S A Pilkington, Principal Investigator — Southampton University
Locations (1):
- Southampton General Hospital, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biofeedback | No Biofeedback
Started | 61 | 60
Completed | 46 | 43
Not Completed | 15 | 17
Not completed — Lost to Follow-up | 9 | 13
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback | No Biofeedback | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10) | 66 (9) | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 38 | 33 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 61 | 60 | 121
Incontinence (CCI) score [Mean (Standard Deviation); unit: scores on a scale] — The Cleveland Clinic incontinence score (CCI) is an anal incontinence severity score. It is easy to use and gives the patient a score of 0 to 20, where zero equates to perfect continence and twenty equates to complete anal incontinence.
  scores on a scale | 4 (5) | 4 (5) | 4 (5)

OUTCOME MEASURES:

1. Primary Outcome: Cleveland Clinic Incontinence (CCI) Score
Description: The Cleveland Clinic incontinence score (CCI) is an anal incontinence severity score. It is easy to use and gives the patient a score of 0 to 20, where zero equates to perfect continence and twenty equates to complete anal incontinence.
Time Frame: 1 year
Population: Analyzed participants, less than the randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biofeedback | No Biofeedback
Number analyzed (Participants) | 43 | 46
score on a scale
  CCI final | 4.2 (4.2) | 3.7 (3.5)
  Adjusted CCI final | 1.2 (6.0) | -0.7 (5.5)
Statistical Analysis 1: Comparison: Biofeedback vs No Biofeedback; CCI final; Test type: Superiority; p = 0.54, Regression, Linear

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Biofeedback | No Biofeedback
All-Cause Mortality (participants affected / at risk) | 1/61 | 4/60
Serious Adverse Events (participants affected / at risk) | 5/61 | 7/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biofeedback (N=61) | No Biofeedback (N=60)
Abdominoperineal excision (Surgical and medical procedures) | 2 (2) | 2 (2)
Hartman procedures (Surgical and medical procedures) | 3 (3) | 4 (4)
Rectovaginal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes